CLINICAL TRIAL: NCT01455961
Title: An Epidemiological Registry Study to Evaluate Clinical Practice Treatment in Patients With Bipolar Disorder Treated With Quetiapine XR and/or Quetiapine IR
Brief Title: An Epidemiological Registry Study to Evaluate Clinical Practice Treatment in Patients With Bipolar Disorder
Acronym: REED
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: VD-NS-1101
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Bipolar Disorder
Keywords: Real life setting; Bipolar Disorder; Registry based Data Base Audit
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to describe the treatment pattern and patient characteristics in real life setting in patients with Bipolar disorder treated with Seroquel XR and/or Seroquel IR in Sweden.

DETAILED DESCRIPTION:
An epidemiological registry study to evaluate clinical practice treatment in patients with Bipolar Disorder treated with quetiapine XR and/or quetiapine IR

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of BD.

Exclusion Criteria:

* Patients with a diagnosis of any schizophrenia spectrum disorder after the diagnosis of bipolar disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have been hospitalised in Sweden at least once since 1987 with a diagnosis during hospitalisation of Bipolar Disorder.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Description of detailed clinical treatment in terms of duration of treatment, doses, drug switches, and add-on therapy, in patients with BD and on treatment with quetiapine XR and/or quetiapine IR before, at and after the index date. | 1st of January 2009 to 31st of December 2010.

SECONDARY OUTCOMES:
Description of co-morbidity, demographics, sick leave, early retirement and socioeconomic factors in patients with BD and on treatment with quetiapine XR and/or quetiapine IR before and at the index date. | 1st of January 2009 to 31st of December 2010.
Description of the detailed clinical treatment in terms of duration of treatment, doses, drug switches, and add-on therapy, in patients with BD, including all drug treatment after the index date | 1st of January 2009 to 31st of December 2010.
Description of co-morbidity, demographics, sick leave, early retirement and socioeconomic factors in patients with BD, including all drug treatment before and at the index date | 1st of January 2009 to 31st of December 2010.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Carlborg, MD, Principal Investigator — Department of Clinical Neuroscience, Karolinska Institutet 171 76 Stockholm

REFERENCES:
- [Derived] Carlborg A, Thuresson M, Ferntoft L, Bodegard J. Characteristics of bipolar disorder patients treated with immediate- and extended-release quetiapine in a real clinical setting: a longitudinal, cohort study of 1761 patients. Ther Adv Psychopharmacol. 2015 Feb;5(1):13-21. doi: 10.1177/2045125314560740. PMID 25653826
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1139&filename=CSR-VD-NS-1101.pdf
- See also: Redacted_protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1139&filename=REED_NCT01455961_Redacted_protocol.pdf